CLINICAL TRIAL: NCT06755008
Title: Benefits of Epithelial Repair in COPD by Induced Pluripotent Stem Cells (iPS)
Acronym: RepCOPDiPS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: MebBioMed (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL24_0012
Record Dates: First submitted 2024-12-05; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; bronchial epithelium; iPS; repair; Club cell
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Interventional, cross-sectional and pathophysiological experimental study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- smoker with COPD (Experimental): Bronchial biopsy performed during a planned bronchial fibroscopy as part of their disease management.
  Interventions: Procedure: bronchial fibroscopy
- smoker without COPD (Active Comparator): Bronchial biopsy performed during a planned bronchial fibroscopy as part of their disease management.
  Interventions: Procedure: bronchial fibroscopy
- healthy non-smoking subject (Active Comparator): Bronchial biopsy performed during a planned bronchial fibroscopy as part of their disease management.
  Interventions: Procedure: bronchial fibroscopy

INTERVENTIONS:
Procedure: bronchial fibroscopy — 2 bronchial biopsies will be taken during bronchial fibroscopy

SUMMARY:
The aim of this interventional, cross-sectional and pathophysiological experimental study is to evaluate the potential of a patient's induced pluripotent stem (iPS) cells, used prior to the re-differentiation stage, to enable ex vivo repair of the injured epithelium in patients with chronic obstructive pulmonary disease (COPD), smokers without COPD and non-smoking controls.

The main questions it aims to answer are:

* to evaluate the repair capacity of bronchial epithelium in COPD subjects, using a model of bronchial epithelium reconstituted in air/liquid interface culture and the iPS model.
* epithelia repair capacities in normal or aberrant situations, as well as the time required for this repair, and to determine the involvement of grafted iPS cells in epithelia repair in cultured control subjects, smokers without COPD and COPD patients.

Researchers will compare 3 groups of participants (COPD patients, smokers without COPD and non-smokers without COPD) for epithelial repair efficacy between non-grafted ALI cultures and ALI cultures grafted with iPS cells, in order to assess their contribution to epithelial repair.

Participants will undergo a bronchial fibroscopy (for clinical indications) with two additional biopsies specific to the study.

This research could lead to breakthroughs in cell-based therapies for COPD, with long-term implications for epigenetic treatments and in vivo applications.

DETAILED DESCRIPTION:
Recently, the research team were able to show that there is a deficiency in a particular subtype of club cells destined to become ciliated in COPD, which would explain the inversion of the ciliated cell/caliciform cell ratio and therefore in the formation of the mucous plugs involved in bronchiolar obstruction.

iPS (induced pluripotent stem cells) represent a major biological breakthrough that has been awarded a Nobel Prize. They offer the advantage of being pluripotent, capable of multiplying endlessly, and thus of differentiating into any other cell type, or even organ, in short, embryogenesis. Researchers have developed a protocol for differentiating iPS cells into bronchial epithelia, with interesting success. These epithelia reconstituted in an air-liquid interface (iALI) reproduce all the characteristics of epithelia in vivo, in particular with the presence of all cell subtypes.

The research team hypothesizes that a patient's iPS cells, used before the re-differentiation stage, will enable ex vivo repair of his damaged epithelium.

The expected results of this project will be to validate the in vitro model of epithelial cell aggression in air-liquid interface (ALI) cultures, and to determine the feasibility of seeding iPS-derived epithelial cells. ALI epithelia from COPD patients would repair better or even normally thanks to iPS.

Ultimately, this project could be a potential therapy targeting epigenetics, and why not a cell therapy.

ELIGIBILITY:
General Inclusion Criteria

* Male and female participants aged 18 years or older.
* Participants with a bronchoscopy indication determined by a pulmonologist (e.g., follow-up exploration, nodule investigation, hemoptysis, cough, sputum production, recurrent bronchitis, or differential diagnosis).

Group 1 Inclusion Criteria: COPD

* Current or former smokers (≥10 pack-years).
* Diagnosed with COPD: FEV1/FVC < 0.7 (confirmed by spirometry available in the medical file within the past year).

Group 2 Inclusion Criteria: Smokers without COPD (n=10)

* Current or former smokers (≥10 pack-years).
* No obstructive ventilatory disorder identified by clinical examination and/or (FEV1/FVC > 0.7 and FEV1 > 70% of predicted values) confirmed by spirometry within the past year.

Group 3 Inclusion Criteria: Non-smoker controls (n=10)

* Never-smokers or former smokers who quit more than 10 years ago (<10 pack-years).
* No obstructive ventilatory disorder identified by clinical examination and/or (FEV1/FVC > 0.7 and FEV1 > 70% of predicted values) confirmed by spirometry within the past year.

Exclusion Criteria:

* Participant with extensive neoplastic disease.
* Participant with another progressive pulmonary condition (e.g., asthma, tuberculosis, interstitial lung disease, active or recent pulmonary infection).
* Participant consuming illicit drugs or alcohol.
* Individual deprived of liberty (by judicial or administrative decision, or under involuntary hospitalization).
* Individual currently enrolled in another research study with an ongoing exclusion period.
* Participant with recent psychiatric disorders (e.g., involuntary hospitalization, mental health conditions preventing informed consent, or requiring immediate medical intervention).
* Adult under legal protection (e.g., guardianship, curatorship, or judicial protection).
* Participant unable to provide informed consent.
* Participant not fluent in French and without a trusted person to assist with comprehension.
* Participant not affiliated with or covered by a social security system.
* Pregnant or breastfeeding women.
* Participant refusing to provide consent after being informed.
* Participant unable or incapable of expressing consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
The main objective is to evaluate the repair capacity of the bronchial epithelium of COPD subjects using the reconstituted bronchial epithelium model in air/liquid interface culture and the iPS model. | Day 1
  Percentage of repair at 24 hours post-lesion of ALI cultures vs. the same ALI cultures "grafted with iPS". This percentage will be determined by the surface area of the culture reconstructed after scratching divided by the surface area initially scratched.

SECONDARY OUTCOMES:
comparison of % repair of post-scratch cultures in the presence or absence of IPS between the 3 groups | Day 2, Day 3 and day 7
  Calculation of the percentage of repair at 48 hours, 72 hours and at 7 days post-scratch. This percentage will be determined by the surface area of the culture rebuilt after scratching divided by the surface area initially scratched.
Comparison of transepithelial electrical resistances between groups | Day 2, Day 3 and day 7
  Verification of the integrity of the bronchial epithelium obtained by measuring the transepithelial electrical resistance. (expressed as Ω/cm2 at each time point).
Determining the proportion of GFP-tagged iPS cells vs. native cells in lesion repair: | Day 2, Day 3 and day 7
  Cell density measurements (% GFP cells/total cells) by microscopy at each time point
Phenotyping of native and GFP+ iPS populations by immunofluorescent labeling of different cell types (ciliated cells, mucus cells, club cells, basal cells) | Day 2, Day 3 and day 7
  immunofluorescence will be used to assess the density of basal, club, ciliated and caliciform cells; the release of key proinflammatory cytokines classically implicated in COPD will be assayed in the supernatant of these cultures.
Comparison of the transcriptomic profile for each cell subtype obtained after sorting native cells and GFP+ iPS cells by flow cytometry. | Day 2, Day 3 and day 7
  Comparison of the transcriptomic profile by ANOVA analysis of the 10 most highly expressed genes between native cells and IPS cells.
Comparison of transcriptomic profile between ungrafted and grafted ALI. | Day 2, Day 3 and day 7
  Comparison of the transcriptomic profile by ANOVA analysis of the 10 most highly expressed genes
ciliated cell/caliciform ratio to check whether the deficient club cell subtype is restored by this technique | Day 2, Day 3 and day 7
  the ciliated cell/caliciform ratio

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde VOLPATO, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- University Hospital of Montpellier, Arnaud de Villeneuve Hospital, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: Undecided